CLINICAL TRIAL: NCT02022917
Title: A Phase II Trial of Postoperative Platinum-based Chemotherapy Plus Adjuvant and Maintenance Bevacizumab After Neoadjuvant Chemotherapy Followed by Interval Surgery in Patients With Extensive Stage IIIC or IV Ovarian, Tubal, and Peritoneal Cancer
Brief Title: Postoperative Adjuvant Chemotherapy With Bevacizumab and Maintenance Bevacizumab After Neoadjuvant Chemotherapy for Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry); Asian Gynecologic Oncology Group (Other); Taiwanese Gynecolgic Oncology Group (Unknown)
Responsible Party: Principal Investigator, Chyong-Huey Lai, M.D., Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGOG11-003; TGOG3008 (Other: Taiwanese GOG)
Record Dates: First submitted 2013-12-11; First posted 2013-12-30 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Epithelial Ovarian Cancer
Keywords: ovarian cancer.; tubal cancer; peritoneal cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epithelial Ovarian Cancer (Experimental): Neoadjuvant Carboplatin, Paclitaxel, and Bevacizumab 21 day cycles of carboplatin, paclitaxel, and bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 15 mg/ Kg (from post-op cycle 2) intravenous infusion for 30 minutes in a 21 days' cycle for at least three cycles (best to 6 cycles) followed by 3-weekly maintenance bevacizumab 15 mg/ Kg intravenous infusion for 17 cycles.
  Other Names: Avastin

SUMMARY:
This study is to determine the feasibility of postoperative platinum-based chemotherapy plus adjuvant and maintenance bevacizumab after neoadjuvant chemotherapy followed by interval surgery in patients with extensive stage IIIC or IV ovarian, tubal, and peritoneal cancer.

DETAILED DESCRIPTION:
This study is designed to determine the feasibility of administering adjuvant carboplatin, paclitaxel, and bevacizumab without unacceptable significant AE in patients with epithelial ovarian cancer after neoadjuvant carboplatin/cisplatin, and paclitaxel and interval cytoreductive surgery, primary peritoneal cancer or fallopian tube cancer. This study will also investigate progression free and to assess the quality of life.

A Simon minimax two-stage design is employed to determine permit early stopping when a moderately long sequence of initial adverse events occurs. Under this two-stage design, 13 subjects are enrolled at the first stage. If there are > 3 subjects discontinue treatment due to significant AE in the stage-1, then stop the trial. Otherwise, the second stage is implemented by including the other 14 subjects. The treatment safety will be evaluated and ensured by the occurrence rate of significant AE (or non AE). In stage-1, postoperative adjuvant cycles 2-6 will be observed for defined significant AE.

Patients' or physicians' decision of discontinuation not because of the above-defined significant AEs or due to cancer progression should not be counted as an end-point event.

ELIGIBILITY:
Inclusion Criteria:

1. previously untreated histologically proven epithelial ovarian cancer, tubal or peritoneal primary carcinoma, of FIGO stage IV or extensive stage III deem not feasible for primary cytoreductive surgery
2. histologic epithelial cell types as follows: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.).
3. well informed about the rationale of neoadjuvant chemotherapy as an alternative to upfront surgery followed by adjuvant chemotherapy and accepted treatment with three to four cycles of neoadjuvant treatment with three to four cycles of platinum-based regimen without progression followed by interval cytoreductive surgery
4. performance status of ECOG 0-2
5. adequate hematopoietic function is defined as below:

   * ANC ≥ 1,500/uL, equivalent to Common Toxicity Criteria for Adverse Events v4.03 (CTCAE) Grade1.
   * Platelets ≥ 100,000/uL (CTCAE Grade 0-1).
   * INR is ≦ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and aPTT < 1.2 x ULN
6. adequate organ function is defined as below:

   * total bilirubin ≦ 1.5 × ULN (CTCAE Grade 1).
   * ALT/AST≦2.5 x ULN and alkaline phosphatase≦2.5 x ULN (CTCAE Grade 1)
   * serum creatinine ≦ 1.5 × ULN (CTCAE Grade 1).
7. adequate neurologic function, neuropathy (sensory and motor) ≦ CTCAE Grade 1
8. age 20-75 years old
9. Patients must have measurable and non-measurable disease. Patients may or may not have cancer-related symptoms.
10. life expectancy equal or longer than 3 months
11. Patients who have met the pre-entry requirements
12. ability to understand and willingness to sign a written informed consent document (within 3 weeks after interval surgery)

Exclusion Criteria

1. borderline ovarian tumors, recurrent epithelial ovarian, tubal or peritoneal or non-epithelial cancers
2. history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarrachnoid hemorrhage within six months of the first date of treatment on this study.
3. Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded.
4. other malignancy with exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to entering the study
5. patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their ovarian, peritoneal primary or fallopian tube carcinoma
6. patients with serious, non-healing wound, ulcer, or bone fracture.
7. patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations.
8. history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months.
9. patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
10. clinically significant proteinuria. Urine protein should be screened by urine protein-creatinine ratio (UPCR). The UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection. Specifically, a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24 hour urine collection. Obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24 hour urine). Send sample to lab with request for urine protein and creatinine levels [separate requests]. The lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL) The UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL). Patients must have a UPCR < 1.0 to allow participation in the study.
11. clinical significant cardiovascular disease

    * Uncontrolled hypertension, defined as systolic >150 mm Hg or diastolic> 90 mm Hg.
    * Prior history of hypertensive crisis or hypertensive encephalopathy
    * active cardiac disease e.g. decompensated myocardial infarction within the 6-month period preceding entry into the study.
    * New York Heart Association (NYHA) Grade II or greater congestive heart failure
    * serious cardiac arrhythmia requiring medication.
    * CTCAE Grade 2 or greater peripheral vascular disease (at least brief (24 hrs) episodes of ischemia managed non-surgically and without permanent deficit)
    * History of CVA within six months.
12. known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
13. presence of other serious concomitant illness which can affect or elevate the value of CA-125, e.g.;

    * Autoimmune disease
    * Sarcoidosis
    * Chronic active hepatitis
    * Pericarditis
    * Cirrhosis of liver
    * Abdominal tuberculosis
    * Pancreatitis
14. acute hepatitis or active infection that requires parenteral antibiotics
15. anticipation of invasive procedures as defined below:

    * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of Bevacizumab therapy (cycle 2).
    * Major surgical procedure anticipated during the course of the study.
    * Core biopsy within 7 days prior to the first date of Bevacizumab therapy (cycle 2).
16. Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
17. concurrent chemotherapy, radiotherapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period
18. mental status is not fit for clinical trial
19. Patients who are pregnant or nursing. Subjects of child-bearing age have to use effective means of contraception
20. Patients who have received prior therapy with any anti-VEGF drug, including bevacizumab.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Significant event rate of the regimen (neoadjuvant carboplatin, paclitaxel, and bevacizumab) | Up to 30 days after the last treatment
  Significant AEs include:
  1. Hypertension ≥ grade 3
  2. Proteinuria ≥ grade 3
  3. GI perforation, abscesses and fistulae (any grade)
  4. Wound healing complications ≥ grade 3
  5. Haemorrhage ≥ grade 3 (any grade CNS bleeding; ≥ grade 2 haemoptysis)
  6. Arterial thromboembolic events (any grade)
  7. Venous thromboembolic events ≥ grade 3
  8. PRES (any grade)
  9. CHF ≥ grade 3
  10. Non-GI fistula or abscess ≥ grade 2

SECONDARY OUTCOMES:
Progression free survival (PFS) | Every 3 months during treatment and every 6 months for three years post-treatment
  Following disease progression, the patient will be contacted every 26 weeks (+/- 2 weeks) (until 30 days after the last patient receives the last dose of bevacizumab) in order to capture their survival status

CONTACTS AND LOCATIONS:
Overall Officials: Chyong-Huey Lai, MD, Study Chair — Chang Gung Memorial Hospital
Locations (5):
- Taiwan (5):
  - Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital, Chiayi City
  - Department of Obstetrics & Gynecology Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Wan Fang Hospital, Taipei Medical University,, Taipei
  - Division of Gynecologic Oncology, Department of Obstetrics & Gynecology Chang Gung Memorial Hospital, Linkou Medical Center, Taoyuan District